CLINICAL TRIAL: NCT00925457
Title: Evaluating the Risk of Serious Ventricular Arrhythmia and Sudden Cardiac Death Among Users of Domperidone
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR016396
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Arrhythmias, Cardiac
Keywords: Serious ventricular arrhythmia; Sudden cardiac death; Domperidone; Case-control study; Saskatchewan residents; Observational Study
MeSH Terms: conditions — Arrhythmias, Cardiac; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- 001: Current Domperidone Current domperidone at any dose regardless of proton pump inhibitor status
  Interventions: Drug: Current Domperidone
- 002: Current proton pump inhibitor (PPI) Current PPI and not current dapoxetine
  Interventions: Drug: Current proton pump inhibitor (PPI)
- 003: No Intervention Neither current domperidone nor current PPI
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Neither current domperidone nor current PPI
  Groups: 003
Drug: Current Domperidone — Current domperidone at any dose, regardless of proton pump inhibitor status
  Groups: 001
Drug: Current proton pump inhibitor (PPI) — Current PPI and not current dapoxetine
  Groups: 002

SUMMARY:
The purpose of this retrospective observational study is to obtain information to confirm or contradict the results of prior studies on domperidone and sudden cardiac death. The population studied are the Saskatchewan residents who used domperidone or another type of medication known as a Proton Pump Inhibitor (PPI) between 1990 and 2005. Information will be collected from various sources including the Saskatchewan Health (SH) database and Cancer Registry.

DETAILED DESCRIPTION:
The purpose of this population-based, observational study is to evaluate the combined risk of serious ventricular arrhythmia (irregular heart rhythm) and sudden cardiac death in users of domperidone (a medication used to treat certain gastrointestinal disorders) compared with users of proton pump inhibitors (another group of medications used to reduce gastric or stomach acid production. The study will be conducted using patient information from Saskatchewan Health (SH) who had recorded dispensings of domperidone or a PPI from 1990 through 2005. The first objective of the study is to estimate the combined relative risk of the occurrence of a particular type of irregular heart rhythm known as serious ventricular arrhythmia (SVA) and sudden cardiac death SCD (defined as a natural death from an unexpected circulatory arrest) during current use of domperidone or current use of proton pump inhibitors (PPIs) as compared with nonuse in a diabetic population. The second objective is to estimate the combined relative risk of SVA and SCD during current use of domperidone or current use of PPIs as compared with nonuse in a non-diabetic population. Study drug dosing information not required for Observational Study

ELIGIBILITY:
Inclusion Criteria:

* Saskachewan residents who received domperidone or a proton pump inhibitor (PPI) between January 1, 1990, and December 31, 2005

Exclusion Criteria:

* Cancer free >=1 year of history in the database before receiving the first dose of domperidone or a PPI

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Saskachewan residents who received domperidone or a proton pump inhibitor (PPI) between January 1, 1990, and December 31, 2005
Sampling Method: Probability Sample
Enrollment: 1608 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The occurrence of serious ventricular arrhythmia and sudden cardiac death (combined end point) | Retrospective study

SECONDARY OUTCOMES:
The second objective is to estimate the combined relative risk of SVA and SCD during current use of domperidone or current use of PPIs as compared with nonuse in a non-diabetic population. | Retrospective

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: Evaluating the Risk of Serious Ventricular Arrhythmia and Sudden Cardiac Death Among Users of Domperidone — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=811&filename=CR016396_Executive_Summary.pdf